CLINICAL TRIAL: NCT01297166
Title: A Psoriasis Plaque Test on LEO 27989 Ointment and Calcipotriol Plus LEO 27989 Ointment in Patients With Psoriasis Vulgaris.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PLQ-006; 2010-022663-35
Record Dates: First submitted 2011-02-03; First posted 2011-02-16 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2013-10

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — calcipotriene

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- LEO 27989 ointment (Experimental)
  Interventions: Drug: LEO 27989 ointment; Drug: Calcipotriol plus LEO 27989 ointment; Drug: Calcipotriol ointment; Drug: Vehicle ointment

INTERVENTIONS:
Drug: LEO 27989 ointment — once daily application, 3weeks
Drug: Calcipotriol plus LEO 27989 ointment — once daily application, 3weeks
Drug: Calcipotriol ointment — once daily application, 3weeks
Drug: Vehicle ointment — once daily application, 3weeks

SUMMARY:
The purpose of this study is to evaluate the anti-psoriatic effect of LEO 27989 ointment and calcipotriol plus LEO 27989 ointment, using the psoriasis plaque test modified from the method developed by KJ Dumas and JR Scholtz.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having understood and signed an informed consent form
* Age 18 years or above
* Males, or females of non-child bearing potential
* All skin types
* Subjects with a diagnosis of psoriasis vulgaris with lesions located on arms and/or legs and/or trunk.

Exclusion criteria:

* Male who are not willing to use a local contraception (such as condom) for the entire duration of the study, and refrain from fathering a child within 3 months following the last study drug application
* Females who are pregnant, of child-bearing potential and who wish to become pregnant during the study, or who are breast feeding
* Systemic treatment with biological therapies (marketed or not marketed) with a possible effect on psoriasis vulgaris within 4 weeks (etanercept), 2 months (adalimumab, alefacept, infliximab), 4 months (ustekinumab) or 4 weeks /5 half-lives (which-ever is longer) for experimental biological products prior to randomisation and during the study
* Systemic treatments with all other therapies than biologicals, with a potential effect on psoriasis vulgaris (e.g., corticosteroids, retinoids, immunosuppressants) within the 4-week period prior to randomisation and during the study
* Subjects using one of the following topical drugs for the treatment of psoriasis within the 4 week period prior to randomisation and during the study:

  * Potent or very potent (WHO group III-IV) corticosteroids
  * PUVA or Grenz ray therapy
* Subjects using one of the following topical drugs for the treatment of psoriasis within two weeks prior to randomisation and during the study:

  * WHO group I-II corticosteroids (except if used for treatment of scalp and/or facial psoriasis)
  * Topical retinoids
  * Vitamin D analogues
  * Topical immunomodulators (e.g. macrolides)
  * Anthracen derivatives
  * Tar
  * Salicylic acid
  * UVB therapy
* Subjects using emollients on the target plaques within one week before randomisation and during the study
* Initiation of, or expected changes to concomitant medication that may affect psoriasis vulgaris (e.g., beta blockers, anti-malaria drugs, lithium and ACE inhibitors) within 2 weeks prior to the randomisation and during the study
* Subjects with current diagnosis of guttate, erythrodermic, exfoliative or pustular psoriasis
* Subjects with known/suspected disorders of calcium metabolism associated with hypercalcaemia based on medical history
* Subjects with a positive Hepatitis B, Hepatitis C or HIV test
* Subjects who have received treatment with any non-marketed drug substance (i.e., an agent which has not yet been made available for clinical use following registration) within the 4 week period prior to randomisation or longer, if the class of the substance requires a longer washout as defined above (e.g., biological treatments)
* Subjects with current participation in any other interventional clinical, based on interview of the subject
* Subjects with known or suspected hypersensitivity to component(s) of the investigational products
* History of any severe disease or serious current condition (based on subject interview and/or results of screening physical examination) which, in the opinion of the Investigator, would put the subject at risk by participating in the study or would interfere significantly with the evaluation of study results or the study course (e.g. cancer, severe cardiopathy, severe renal insufficiency, severe hepatic insufficiency).
* Subjects with a positive Hepatitis B, Hepatitis C or HIV test
* Subjects with any concomitant medical or dermatological disorder(s) which might preclude accurate evaluation of the psoriasis on the test areas
* Subjects foreseeing an intensive solar exposure during the study (UV radiation, etc.) or having been exposed within two weeks preceding the screening visit
* Subjects with any contraindication to skin biopsy procedures: e.g., allergy to local anaesthetics, topical antiseptics (chlorhexidine), bleeding tendency, treatment with anticoagulant drugs, history of poor wound healing, and history of vasovagal hypotension or syncope.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Absolute change in Total Clinical Score (TCS) of clinical symptoms (sum of erythema, scaling and infiltration) at end of treatment compared to baseline. | 3 weeks
  TCS range from 0 (all symptoms absent) to 9 (all symptoms severe)

SECONDARY OUTCOMES:
Clinical sympton scores | 3 weeks
  Absolute change in single clinical symptom score: erythema, scaling, infiltration at end of treatment and individual visits compared to baseline.
  Change in Total Clinical Score (TCS) at individual visits compared to baseline.
Lesion thickness | 3 weeks
  Change in lesion thickness measured by ultrasound at each assessment compared to baseline.
Immunohistochemical and histologic scoring of biopsy material | 3 weeks
Intra-subject variability | 3 weeks
  The intra-subject variability of changes from baseline to end of treatment of TCS and skin thickness

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Queille-Roussel, MD, Principal Investigator — Centre de Pharmacologie Clinique Applique a la Dermatologie
Locations (1):
- CPCAD, Nice, France

IPD SHARING:
Plan to Share IPD: No